CLINICAL TRIAL: NCT00586846
Title: Phase II Study of Chemotherapy and Pamidronate for the Treatment of Newly Diagnosed Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-074; NCT00072306 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Osteosarcoma
Keywords: Cisplatin; Doxorubicin; Methotrexate; Osteosarcoma; 03-074
MeSH Terms: conditions — Osteosarcoma | interventions — Cisplatin; Doxorubicin; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Cisplatin; Drug: Doxorubicin; Drug: Methotrexate

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 120 mg/m^2
Drug: Doxorubicin — 75mg/m^2
Drug: Methotrexate — Methotrexate 12g/m^2

SUMMARY:
This study is designed to test the safety and feasibility of the simultaneous administration of a biphosphonate with chemotherapy for the treatment of osteosarcoma in newly diagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated biopsy proven high-grade osteosarcoma. Patient who have undergone a definitive surgical resection as their primary surgery are still eligible for participation in this study.
* No prior chemotherapy or radiation therapy
* Adequate renal function: creatinine < or = to 1.5 upper limit of normal
* Adequate liver function as defined by bilirubin < or = to 1.5 X upper limit of normal and AST < or = to 3 X upper limit of normal institutional range Adequate hematopoietic function as defined by platelet count > or = to 100,000/ram3 an absolute neutrophil count > or = to 1,000/mm3.
* Adequate cardiac function as defined by shortening fraction > or = to 28% by echocardiogram OR ejection fraction > or = to 50% by radionuclide angiogram
* Performance status < or = to 2

Exclusion Criteria:

* Prior history of cancer
* Prior treatment for cancer
* Prior history of Paget's disease
* Prior history of pericarditis, myocarditis, symptomatic arrhythmia or symptomatic cardiac conduction abnormalities
* Pregnancy or breast feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meyers Paul, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Chemotherapy and Pamidronate for the Treatment of Newly Diagnosed Osteosarcoma
Period: Overall Study
Arm/Group | All Patients
Started | 40
Completed | 34
Not Completed | 6
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Evaluable for Toxicity Only | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response
Description: to the induction chemotherapy in the primary tumor and in any metastatic lesions using the Response Evaluation Criteria (RECIST).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 34
participants
  Complete Response (CR) | 21
  Partial Response (PR) | 5
  Stable Disease (SD) | 5
  Progression of Disease (POD) | 3

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 25/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=40)
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Febrile neutropenia (General disorders) | 4 (9)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 1 (2)
Intraoperative reproductive tract (Reproductive system and breast disorders) | 1 (1)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 2 (2)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 4 (4)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=40)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 17 (17)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
ALT, SGPT (Metabolism and nutrition disorders) | 37 (37)
Anorexia (General disorders) | 8 (8)
AST, SGOT (Metabolism and nutrition disorders) | 37 (37)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 19 (19)
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 16 (16)
Constipation (Gastrointestinal disorders) | 7 (7)
Dehydration (Gastrointestinal disorders) | 2 (2)
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 4 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4)
Febrile neutropenia (General disorders) | 25 (25)
Fever (in the absence of neutropenia) (General disorders) | 7 (7)
Flushing (Skin and subcutaneous tissue disorders) | 3 (3)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 39 (39)
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 6 (6)
Hair loss/alopecia (scalp or body) (General disorders) | 14 (14)
Hemoglobin (Blood and lymphatic system disorders) | 40 (40)
Hemorrhage, Nose (General disorders) | 4 (4)
Hypertension (Cardiac disorders) | 2 (2)
Catheter Related Infection (Infections and infestations) | 6 (9)
Infection, other (Infections and infestations) | 2 (2)
International Normalized Ratio (INR) (Blood and lymphatic system disorders) | 3 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 40 (40)
Lymphopenia (Blood and lymphatic system disorders) | 33 (33)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 17 (17)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 4 (4)
Mucositis (Clincal exam)- Oral cavity (General disorders) | 23 (23)
Mucositis (Clincal exam)- Pharynx (General disorders) | 3 (3)
Mucositis (symptoms)- Oral cavity (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 19 (19)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 40 (40)
Pain - Abdomen NOS (General disorders) | 2 (2)
Pain - Back (General disorders) | 2 (2)
Pain - Dental/teeth/peridontal (General disorders) | 2 (2)
Pain - Extremity-limb (General disorders) | 7 (7)
Pain - Head/headache (General disorders) | 2 (2)
Pain - Other (General disorders) | 10 (10)
Pain - Throat/pharynx/larynx (General disorders) | 2 (2)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 38 (38)
Platelets (Blood and lymphatic system disorders) | 39 (39)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 13 (13)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 17 (17)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 12 (12)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 18 (18)
Tinnitus (General disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes